CLINICAL TRIAL: NCT04485910
Title: Sequential Versus Single Step Culture Media in Relation to Euploidy Rates in PGTai Program
Brief Title: PGTai Results for Embryos Cultured in Sequential Versus Single Step Media
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MH0004
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Infertility; Aneuploidy Rate; Mosaicism
Keywords: PGT-A; Mosaicism; Single step media; Sequential media
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Evaluating the embryonic development and PGTai results for embryos cultured in sequential media versus single step media.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single step media (Active Comparator): Embryos cultured in single step media
  Interventions: Other: Single step media
- Sequential media (Active Comparator): Embryos cultured in sequential media
  Interventions: Other: Sequential media

INTERVENTIONS:
Other: Single step media — Usage of single step media in embryo culture
  Arms: Single step media
Other: Sequential media — Usage of sequential media in embryo culture
  Arms: Sequential media

SUMMARY:
A prospective cohort study undergoing ICSI at a private fertility center in Egypt

DETAILED DESCRIPTION:
Purpose:

To evaluate PGTai results for embryos cultured in sequential versus single step media.

Method:

Injected oocytes will divided between Continuous Single Culture-NX media (CSC- NX) with 10% SSS the first group (Irvine, USA) and the other group will be cultured in sequential cleavage and blastocyst media with 10% SPS (SAGE, Denmark).

All blastocytes with 4BB quality and better according to Gardner's criteria 1999 will go through PGTA procedures with PGTai confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≤37 years with ≥ 8 mature oocytes
* Male partner had normal semen parameters according to WHO 2010
* PGT-A was done at the blastocyst stage

Exclusion Criteria:

* sperm or oocyte donor
* severe male factors according to WHO 2010

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female age ≤37 years with ≥ 8 mature oocytes
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Euploidy rate | 5:7 days of intracytoplasmic sperm injection(ICSI)
  percentage of euploid embryos/ total genetic tested embryos on blast stage
Mosaicism rate | 5:7 days of ICSI
  percentage of mosaic embryos/ total genetic tested embryos on blast stage

SECONDARY OUTCOMES:
Fertilization rate | 16:19 hours of ICSI
  Percentage of fertilized oocyte (appearance of two pronuclei) / Number of injected oocytes
Cleavage stage | 72 hours of ICSI
  Percentage of cleaved embryos/ total number of fertilized oocytes
High quality of cleaved embryos | 72 hours of ICSI
  High quality D3 embryos according to Gardner's criteria / total cleaved embryos
Blast formation rate | 5:7 days of ICSI
  Percentage of total blastocysts / Total cleaved embryos
High quality blast rate | 5:7 days of ICSI
  Morphological grading of trophectoderm and Inner cell mass using Gardner's criteria 1999, from grade A and B ( A is the highest quality). Total high grade embryos/ total blast embryos.

CONTACTS AND LOCATIONS:
Overall Officials: Manar M Hozyen, MSc., Principal Investigator — Ganin Fertility Center; Amr Elshimy, BSc., Principal Investigator — Ganin Fertility Center; Hanaa Elkhader, BSc., Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc., Study Chair — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Egypt